CLINICAL TRIAL: NCT06451796
Title: A Urethral Valve Catheter for the Treatment of Women With Stress Urinary Incontinence (SUI)
Brief Title: Investigation of Novel Non-CE Marked Catheter
Status: Recruiting | Type: Observational
Sponsor: MagCath (Unknown)
Collaborators: Herlev Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CIV-23-10-044313
Record Dates: First submitted 2024-05-28; First posted 2024-06-11 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Female Stress Incontinence
Keywords: Female Stress Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Obtinu — Treatment of Female Stress Incontinence with a hydrophilic coated valved intraurethral catheter

SUMMARY:
Hypothesis: Treatment with the hydrophilic coated valved intraurethral catheter up to 16 hours per day is effective, well tolerated and seemingly safe for treatment of women with stress incontinence.

Test persons: Ten to twenty stress incontinent women. Treatment time: Up to two weeks

DETAILED DESCRIPTION:
Demonstrate ease and comfort of device insertion, indwelling and removal. Patient acceptability during use.

Other:

* Symptom and QOL questionnaire.
* Drop out analysis.
* Is the patient motivated to continue using the valve catheter?
* Is the patient motivated to recommend the valve catheter to other stress incontinent women?

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate
* Adult, competent woman who understands Danish.
* SUI as dominant symptom; daily or almost daily.
* Residual urine < 150 ml.
* POP-Q prolapse ≤ grade 2.
* Negative urine stix/Urine D+R.
* Min. 2 months local vaginal estrogen treatment if the woman is postmenopausal.
* Mobile and self-reliant woman.
* Motivated.

Exclusion Criteria:

* Allergy to the silicone material
* Pregnancy or breastfeeding
* Unexplained hematuria.
* Current inflammatory disorders
* Malignant disorders of the urethra.
* Urethral stricture
* Visual diverticulum.
* AK treatment.
* Prosthetic heart valve surgery.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women suffering from stress urinary incontinence
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Safety primary: Migration of device to bladder | 2 weeks
  Number of Participants with Migration of device to bladder

SECONDARY OUTCOMES:
Safety secondary: Culture confirmed urinary tract infections. | 2 weeks
  Number of Participants with urinary tract infections.
Safety secondary:Need for antibiotics. | 2 weeks
  Number of Participants with need for antibiotics.
Safety secondary: Discomfort at self-catheterization. | 2 weeks
  Number of Participants with discomfort at self-catheterization.
Safety secondary: Difficulties emptying the bladder. | 2 weeks
  Number of Participants with difficulties emptying the bladder.
Safety secondary: Discomfort at catheter removal. | 2 weeks
  Number of Participants with discomfort at catheter removal.
Safety secondary: Hematuria (stick test/macroscopic). | 2 weeks
  Number of Participants with Hematuria (stick test/macroscopic).
Safety secondary: Allergy. | 2 weeks
  Number of Participants with Allergy.
Safety secondary: Loss of device. | 2 weeks
  Number of lost devices

OTHER OUTCOMES:
Functionality: Is long term continuous use acceptable? | 2 weeks
  Is long term continuous use acceptable?

CONTACTS AND LOCATIONS:
Overall Officials: Pia Sander, MD PhD, Principal Investigator — Herlev Hospital
Locations (1):
- GynCare, Herlev, DK, Denmark

IPD SHARING:
Plan to Share IPD: No